CLINICAL TRIAL: NCT03756727
Title: Effect of Perioperative Application of Ascorbic Acid on Postoperative Pulmonary Complications in Patients Undergoing Cardiac Surgery
Brief Title: Effect of Ascorbic Acid on Postoperative Pulmonary Complications in Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Principal Investigator, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XYFY-2018-1101
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pulmonary Complications
MeSH Terms: interventions — Ascorbic Acid; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascorbic acid group (Experimental): the patients received 2g of intravenous Ascorbic acid at the night before surgery, during the surgery and five days after surgery.
  Interventions: Drug: Ascorbic Acid
- Control comparator group (Placebo Comparator): the patients received 10ml saline at the night before surgery, during the surgery and five days after surgery.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ascorbic Acid — Patients in Ascorbic acid group received 2g of intravenous Ascorbic acid at the night before surgery, during the surgery and five days after surgery (once a day).
  Other Names: Vitamin c
  Arms: Ascorbic acid group
Drug: Saline — Patients in Control Comparator group received saline 10ml at the night before surgery, during the surgery and five days after surgery (once a day).
  Other Names: Saline Solution
  Arms: Control comparator group

SUMMARY:
Postoperative pulmonary complications(PPCs) including, but not limited to ,hypoxemia, pneumonia, ventilator-induced lung injury, and acute respiratory distress syndrome (ARDS),atelectasis,pleural effusion .PPCs may result in increased resources utilization, delayed mobilization, prolonged need of supplemental oxygen or mechanical ventilation,and a longer hospital stay.postoperative pulmonary complications are common after cardiac surgery, often increasing postoperative morbidity and mortality.The extracorporeal circulation,increased oxygen concentration inhaled and the development of massive atelectasis after open-chest surgery commonly activate lung inflammation, amplifying the harm Injury of pulmonary .Currently, plenty of interventions have been studied to prevent PPCs after surgery. Most of the recent research has focused on physical therapy such as lung-protective modes during intraoperative mechanical ventilation, Alveolar Recruitment, and respiratory muscle training.These therapies have a certain effect, but still not satisfactory.Ascorbic acid is an important cofactor in multiple enzymatic reactions where its main function is as a reducing agent.Studies have shown that ascorbic acid can reduce both ischemia-reperfusion injury and oxidative stress. Unfortunately, no studies examined whether Ascorbic acid can reduce PPCs.

DETAILED DESCRIPTION:
The possible mechanisms of ascorbic acid to alleviate ischemia-reperfusion injury are as follows: 1 Ascorbic acid as a first-line antioxidant in plasma can reduce stress by eliminating excess Reactive oxygen species and reduce damage. 2 provides rapid electron transfer to react with superoxide and hydroxyl group to scavenge reactive oxygen released into the circulation. 3 Ascorbic acid can reduce lipid peroxidation and reduce lung injury caused by ischemia-reperfusion by scavenging oxygen free radicals. 4 Vitamin C can promote the production of cytokines by immune cells to reduce local inflammatory reactions and improve tissue microcirculation.The study aims to explore whether daily used Ascorbic acid in the perioperative period has a preventive effect on PPCs in patients undergoing cardiac surgery, and through short-term and long-term follow-up, to investigate the effect on post-hospitalization Prognosis .

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60 years old
2. Selective cardiac surgery under cardiopulmonary bypass

Exclusion Criteria:

1. Emergency surgery
2. Previous cardiac surgery
3. Severe lung disease
4. BMI<18 or >30
5. Mean pulmonary arterial pressure >40 mmHg
6. were allergic to ascorbic acid

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
severity of postoperative pulmonary complications | an average of 2 weeks
  Use the postoperative pulmonary complications score to record the severity. scored ranging from 0 to 5.Scored the severity once a day, record the highest score.

SECONDARY OUTCOMES:
incidence of postoperative pulmonary complications | an average of 10 days
  incidence of postoperative pulmonary complications during hospital stay
length of ICU stay and length of hospital stay | an average of 10 days
  all patients transfer to ICU after surgery
extubation and wake time | an average of 1 day
  length of extubation time,length of wake time
PaO2/FiO2 | 1 day, 3 days,5 days post surgery
  Oxygenation index (PaO2/FiO2) in millimeter mercury column.
A-aDO2 | 1 day, 3 days,5 days post surgery
  alveolar-arterial oxygen tension difference (A-aDO2)
Plateau pressure | an average of 1 day
  Plateau pressure in centimeter water column
Peak airway pressure | an average of 1 day
  Peak airway pressure in centimeter water column
positive end expiratory pressure | an average of 1 day
  positive end expiratory pressure in centimeter water column
lung compliance | an average of 1 day
  lung compliance in Milliliter/ centimeter water column
post-hospitalization follow-up | once a day till 30 days post-hospitalization
  record the incidence of postoperative pulmonary complications after hospital discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Dong Liu, M.S, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data(IPD) will be available when this trial is finished and the article have been published

REFERENCES:
- [Background] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Background] Baker WL, Coleman CI. Meta-analysis of ascorbic acid for prevention of postoperative atrial fibrillation after cardiac surgery. Am J Health Syst Pharm. 2016 Dec 15;73(24):2056-2066. doi: 10.2146/ajhp160066. Epub 2016 Nov 2. PMID 27806938
- [Background] Costa Leme A, Hajjar LA, Volpe MS, Fukushima JT, De Santis Santiago RR, Osawa EA, Pinheiro de Almeida J, Gerent AM, Franco RA, Zanetti Feltrim MI, Nozawa E, de Moraes Coimbra VR, de Moraes Ianotti R, Hashizume CS, Kalil Filho R, Auler JO Jr, Jatene FB, Gomes Galas FR, Amato MB. Effect of Intensive vs Moderate Alveolar Recruitment Strategies Added to Lung-Protective Ventilation on Postoperative Pulmonary Complications: A Randomized Clinical Trial. JAMA. 2017 Apr 11;317(14):1422-1432. doi: 10.1001/jama.2017.2297. PMID 28322416